CLINICAL TRIAL: NCT04034316
Title: A Phase 2 Open-label Study to Evaluate the Efficacy of Allogeneic Human Cord Blood-derived Mesenchymal Stromal Cells in Maintaining Remission After Immunosuppressive Therapy Withdrawal in Pediatric Patients With Steroid-dependent Nephrotic Syndrome
Brief Title: Reduce Immunosuppression With Atmp in NS ChildrEn
Acronym: RACE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: Cell Factory Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico (Unknown); Laboratorio Sperimentale di Immunologia e Trapianti, Oncoematologia Pediatrica, Fondazione IRCCS Policlinico S. Matteo, Pavia (Unknown)
Responsible Party: Principal Investigator, Giovanni Montini, Professor, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIFA-2016-02364896; 2018-001162-42 (EudraCT Number)
Record Dates: First submitted 2019-07-25; First posted 2019-07-26 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Nephrotic Syndrome in Children; Steroid-Dependent Nephrotic Syndrome; Idiopathic Nephrotic Syndrome
Keywords: Mesenchymal Stromal Cells; Steroid Dependent Nephrotic Syndrome in Children; Proteinuria; Immunosuppressive treatment
MeSH Terms: conditions — Nephrotic Syndrome; Nephrosis, Lipoid; Proteinuria

STUDY DESIGN:
Intervention Model Description: Open lable, single arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MSC (Experimental): During the first part of the study, 11 SDNS pediatric patients will receive 3 intravenous infusions of CB-MSCs at the dosage of 1.5 x 10^6/kg at a time interval of 1 to 2 weeks. The ongoing immunosuppressive treatment will be gradually tapered off after the first CB-MSC administration, as follows:
  * 25% reduction of the ongoing immunosuppressive treatment following the first administration;
  * 50% reduction of the ongoing immunosuppressive treatment following the second administration;
  * interruption of the ongoing immunosuppressive treatment following the third administration.
  In the case that the hypothesis that P ≥ 0.600 is rejected and therefore the second part of the study will be required, 11 additional pediatric patients with SDNS will be treated with 3 intravenous infusions of CB-MSCs at the dosage of 2x10^6/kg at a time interval of 1 to 2 weeks.
  Interventions: Other: Cord-blood mesenchymal stromal cells

INTERVENTIONS:
Other: Cord-blood mesenchymal stromal cells — The product is packaged in bags suitable for the cryopreservation of cell products. Before administration the cells must be thawed and diluted in an appropriate vol:vol solution: made by saline 78%, human albumin 10%, Acyl-CoA dehydrogenase-A (ACD-A) 12%.

SUMMARY:
A phase II open-label, single arm study aimed to ascertain whether infusions of cord-blood mesenchymal stromal cells (CB-MSCs) allow to reduce or suspend the chronic immunosuppressive therapy (IS) in steroid-dependent nephrotic syndrome (SDNS).

We plan to enroll 11 patients aged 3 to 18 with SDNS in remission for at least one month, maintained by either ≥2 immunosuppressive drugs or a calcineurin inhibitor.

Patients are infused with cord-blood allogenic MSC, selected by in-vitro alloreactivity, at a dose of 1.5x10^6/kg on days 0, 14, 21. The immunosuppressive treatment is gradually tapered starting at the first CB-MSC administration, according to the following scheme: 25% following the first administration, 50% following the second administration, and 100% reduction following the third administration.

All patients will be followed-up for 6 months from the last CB-MSC. Study visits are planned at baseline during CB-MSC administrations, 2 weeks (follow-up [FU]1) and 6 weeks (FU2) after the last infusion, and then every 6 weeks. During follow-up, the patients undergo a physical examination (including measurement of height, weight and blood pressure) and laboratory evaluations (urinary protein:urinary creatinine ratio, complete blood count, kidney function, plasma proteins, liver function, triglycerides and cholesterol). In addition, a blood sample is taken for regulatory T lymphocyte quantification, a marker of clinical response to the infusions.

DETAILED DESCRIPTION:
Background:

Nephrotic Syndrome (NS) is a rare disease characterized by nephrotic-range proteinuria and the need for steroid treatment. About 50% of children will become frequent relapsers (FRNS) or steroid dependent (SDNS), requiring higher doses of steroids or other immunosuppressive drugs for many years, sometimes up to adulthood. Strong evidence suggests that Idiopathic nephrotic syndrome (INS), at least in the steroid-sensitive forms, has an immune pathogenesis.

Mesenchymal Stromal Cells (MSC) are multipotent non-hematopoietic stem cells that produce an immunomodulatory activity in-vitro and in-vivo. For this reason, we postulated that SDNS patients could benefit with treatment with MSC.

Objectives:

The main goal of the present study is to assess whether CB-MSCs have the capacity to regulate the immunologic mechanisms involved in the pathogenesis of NS allowing for a reduction or suspension of chronic immunosuppressive treatment in SDNS children. The primary objective is to evaluate whether CB-MSC therapy is able to prevent NS recurrence for at least 6 months after complete withdrawal of immunosuppressive treatment in children with SDNS.

Primary endpoint: percentage of children without NS recurrence after complete withdrawal of immunosuppressive treatment for at least 6 months.

Population:

We plan to enroll 11 children (3 to 18 years of age) with SDNS, maintained by chronic immunosuppressive treatment and with stable remission for at least two months.

Study Design:

Open label single-arm, monocentric trial, with a rescue/second design

Phase: Phase II

Inclusion/Exclusion Criteria:

Inclusion criteria

1. Age between 3 and 18 years;
2. Clinical diagnosis of SDNS;
3. Disease remission maintained by chronic therapy (at least 6 months) with either:

   * Use of a combination of 2 or more immunosuppressive drugs
   * use of 1 of the calcineurin inhibitors (Cyclosporin or Tacrolimus);
4. Absence of proteinuria (urinary protein:urinary creatinine < 0.2 mg/mg) for at least 1 month;
5. Estimated glomerular filtration rate greater than or equal to 70 ml/min/1.73 m^2;
6. Written informed consent from parents or guardians and the child when possible.

Exclusion criteria

1. Age < 3 years or ≥ 19 years;
2. Resistant/refractory NS;
3. Presence of genetic mutations associated with NS;
4. eGFR less than 70 ml/min/1.73 m^2;
5. Thrombophilic condition;
6. Pregnancy or lactating;
7. Evidence of an uncooperative attitude;
8. Any evidence that the patient will be unable to complete the trial follow-up.

Description of the Intervention:

The trial will rely on a single advanced therapy medicinal product (ATMP), made by MSC from umbilical cord blood (CB) for allogeneic use, produced following a highly standardized process, developed and controlled at Cell Factory under the Good Manufacturing Practices guidelines.

After baseline clinical and laboratory evaluation, patients will receive 3 intravenous infusions of CB-MSCs at the dosage of 1.5 x 10^6/kg at a time interval of 1 to 2 weeks.

The immunosuppressive treatment will be gradually tapered off following the first CB-MSC administration: 25%, 50% and 100% reduction of the ongoing immunosuppressive treatment following the first, second and third administration, respectively.

At the end of this first part of the trial, a statistical analysis will be performed according to the primary end-point. In the case of failure to reach the primary end point an extra 11 children with SDNS will be enrolled in a single stage phase 2 study with a 30% incremented dose of CB-MSCs.

Statistical Evaluation:

A phase II design with a rescue plan B, is adopted to decide whether the proportion responding is less than or equal to 0.200 or greater than or equal to 0.600. A sample size of 10 children is required, considering a drop out of 10%, 11 children will be enrolled: if the number of responses is 5 or more, the hypothesis that P ≤ 0.200 is rejected with a target error rate of 5%. If the number of responses is 4 or less, the hypothesis that P ≥ 0.600 is rejected with a target error rate of 20% (power equal to 80%). The same statistical hypothesis will apply for the second part of the study.

Expected Results:

The results of this proposal will provide information regarding an innovative cell therapy for the treatment of INS. If the hypothesis of this study is confirmed, it will be possible to reduce or withdraw immunosuppressive treatment in this vulnerable population of children with SDNS, reducing the need for ambulatory visits and hospitalization and therapy-related complications. Furthermore, the reduction in the use of immunosuppressive agents as well as in the number of outpatient visits and hospital admissions will reduce the financial burden to the National Health Service. Above all, the quality of life of children with SDNS would clearly be improved, in terms of a reduction in long-term therapy, morbidity and the number of visits.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 3 and 18 years;
2. Clinical diagnosis of SDNS;
3. Disease remission maintained by chronic therapy (at least 6 months) with either:

   * Use of a combination of 2 or more immunosuppressive drugs
   * use of 1 of the calcineurin inhibitors (Cyclosporin or Tacrolimus);
4. Absence of proteinuria (PrU/CrU < 0.2 mg/mg) for at least 1 month;
5. eGFR greater than or equal to 70 ml/min/1.73 m^2;
6. Written informed consent from parents or guardians and the child when possible

Exclusion Criteria:

1. Age < 3 years or > 19 years;
2. Resistant/refractory NS;
3. Presence of genetic mutations associated with NS;
4. eGFR less than 70 ml/min/1.73m2;
5. Thrombophilic condition;
6. Pregnancy or lactating;
7. Evidence of an uncooperative attitude;
8. Any evidence that the patient will be unable to complete the trial follow-up.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
The percentage of patients without nephrotic syndrome recurrence after complete withdrawal of immunosuppressive treatment for at least 6 months | 6 months following completion of the intervention
  The percentage of patients without nephrotic-range proteinuria as measured by the urinary protein to urinary creatinine ratio (uPr/uCr<2) 6 months after completing the intervention

SECONDARY OUTCOMES:
The percentage of adverse events | 6 months following completion of the intervention
  As described by the Common Terminology Criteria for Adverse Events
The time to recurrence of nephrotic syndrome | Within 6 months from the completion of the intervention
  As measured by the ratio of urinary protein to urinary creatinine
The percentage of participants achieving a reduction in the immunosuppressive therapy | 6 months following completion of the intervention
  Reduction of the ongoing immunosuppressive treatment
The dose of immunosuppressive therapy to prevent further NS relapses | 6 months following completion of the intervention
  The minimal dose of immunosuppressive therapy necessary to maintain the patient in remission following the therapy
Reported Quality of Life | 6 months following completion of the intervention
  Changes in quality of life as reported by the patients and/or parents

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Nephrology, Dialysis and Transplant Unit, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico Milan, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Undecided